CLINICAL TRIAL: NCT06765824
Title: Transcranial Magnetic Stimulation in the Treatment of Dual Disorders: Study in Patients with Depression and Tobacco Addiction
Brief Title: Transcranial Magnetic Stimulation in Patients with Dual Disorders
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Cardenal Herrera University (Other)
Collaborators: Hospital Provincial de Castellon (Other)
Responsible Party: Principal Investigator, Gonzalo Rafael Haro Cortés, Medical specialist in Psychiatry. Head of the dual disorders program at the "Hospital Provincial de Castellón". Professor in the Department of Medicine and Surgery at the "Universidad Cardenal Herrera-CEU", CEU Universities., Cardenal Herrera University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CEIm-64-02
Record Dates: First submitted 2024-12-18; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Major Depression; Tobacco Addiction
Keywords: Transcranial Magnetic Stimulation; Major depressive disorder; Tobacco Addiction; Dual disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Intervention Model Description: Patients who meet the inclusion criteria will be randomized into a control group, which will receive the active treatment. The control group will receive placebo.
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Transcranial Magnetic Stimulation-Active Coil (Experimental): Patients in the experimental group will receive transcranial magnetic stimulation treatment using an active coil, cool-B70. The protocol to be administered is composed of 36 sessions that will be divided into two sessions per day, with a 50-minute break between sessions. For three months after the main treatment (protocol described above), a booster dose will be administered once a week.
  Interventions: Device: Repetitive Transcranial Magnetic Stimulation
- Transcranial Magnetic Stimulation-Sham coil (Sham Comparator): The control group will receive the same protocol as the experimental group, with the main difference being that this group receives treatment through a placebo coil, MCF-P-B70. The placebo coil maintains the appearance and sound of the one that administers the active treatment, but differs from this in that it does not generate an effective magnetic field capable of generating depolarization in the stimulated brain area.
  Interventions: Device: Transcranial Magnetic Stimulation Sham

INTERVENTIONS:
Device: Repetitive Transcranial Magnetic Stimulation — The protocol will be applied with the MagVenture R30 stimulation device and the cool-B70 coil for active treatment. The protocol will consist of two sessions per day, with a 50-minute break between sessions, every day of the week (Monday to Friday) for three and a half weeks (a total of 36 sessions). Each session will consist of the application of a 1Hz protocol (2000 pulses at 120% of the motor threshold) in the right dorsolateral prefrontal cortex (F4) followed by an intermittent theta-burst protocol (1800 pulses at 90% of the motor threshold) in the left dorsolateral prefrontal cortex (F3). The cortical target localization will be performed using the beam-F3/F4 technique that combines different electroencephalographic positioning parameters and measurements to accurately locate said cortical targets. The motor threshold of each patient will be calculated at the beginning of each week of treatment using an electromyography system.
  Arms: Transcranial Magnetic Stimulation-Active Coil
Device: Transcranial Magnetic Stimulation Sham — The same protocol described in the intervention group will be carried out in the control group. The device used is the same, the difference is the coil that maintains the same appearance and generates the same sound as the active treatment coil, but unlike the latter, it does not produce an effective magnetization to depolarize the cerebral cortex on which we act.
  Arms: Transcranial Magnetic Stimulation-Sham coil

SUMMARY:
According to the WHO, 280 million people are diagnosed with depression, the prevalence of which is almost twice as high in women as in men, with the incidence among young people increasing in recent years. Another public health problem in Spain is tobacco consumption, with one in four adults being tobacco users. The presence of an addiction and another mental illness in the same patient is called dual disorder, and it is very common for depression to be associated with smoking. This is due to a shared biopsychosocial vulnerability between the two disorders. Although there are currently pharmacological treatments that address both disorders, their efficacy is limited; in this sense, transcranial magnetic stimulation (TMS) offers a way to treat these dual disorders. TMS is a technique in which a magnetic field is applied to the cortex through a coil, generating an electric current that can induce changes in the different neurotransmitter systems, stimulating or inhibiting them. A randomised, double-blind, placebo-controlled clinical trial is proposed to evaluate the efficacy of TMS in the treatment of a sample of 36 patients with resistant major depression and nicotine dependence. Both depression and smoking will be assessed at baseline, at various times during treatment and at the end of the study using psychometric tests, neurophysiological and biochemical assessments. It is expected that the experimental group will show improvements in depression, nicotine dependence and certain cognitive functions. TMS treatment of dual disorders (resistant depression + smoking) could represent a health and social advance, especially for women.

DETAILED DESCRIPTION:
Currently, resistant major depression and substance abuse disorder are two highly prevalent mental health pathologies. In the case of depression, the WHO estimates that 3.8% of the world's population suffers from this disorder, which is the result of a complex interaction between social, biological and psychological factors. Multiple sociodemographic factors are related, such as low socioeconomic status, which results in a poorer physical condition that predisposes to depression. In addition, there is also a strong association with different mental illnesses, when associated with an addiction it is called Dual Disorder, with tobacco or alcohol consumption being more frequent. Other factors to highlight are a history of trauma in childhood, being in a situation of divorce/separation, but there is especially a strong association with the female gender. Although the prevalence in the female gender is much higher, no difference is observed with respect to men in terms of the course of the disease and the risk of relapse. The higher incidence of depression in women can be attributed to different factors: biological reasons (hormones and genetic load), psychological reasons (neuroticism, lack of positive affect, rumination or personal dissatisfaction), without forgetting environmental factors: such as sexual abuse or violence in childhood, as well as social inequalities between men and women. This clear difference between women and men justifies and demands the incorporation of a gender perspective in the research, management and treatment of patients diagnosed with major depression. The importance of major depression also lies in the fact that it is the fourth cause of death in the age group between 15 and 29 years and is a common cause of temporary disability due to common contingencies in people of working age, with durations of around 6 months, much longer than the duration estimated by the National Institute of Social Security of 30-60 days. This is reflected in the economic costs, which are estimated to result in an annual public expenditure of up to 10,763 million euros. It is a complex disease that is expected to see its incidence increase in the coming years, which is why it requires a scientific effort for its diagnosis and treatment, especially in resistant cases, because they evolve into a chronic mental illness with higher personal, social and health costs. Nicotine use disorder is also a public health problem, with 50,000 deaths currently attributed to it. The prevalence of 1 in 4 individuals makes it the most common mental illness. Although there has been a decline in consumption among men in recent years, this is not reflected in the same way among women. There are many factors that determine vulnerability to nicotine use disorder, both genetic and psychosocial, highlighting that the early onset of consumption predisposes to a higher risk of addiction, given the brain immaturity in certain brain circuits. Due to biopsychosocial factors common to other mental disorders, it is common for patients with tobacco addiction to present dual disorder, especially depressive disorders. An example is the CHRNA5 gene, encoding the alpha 5 subunit of the acetylcholine receptor, related to nicotine dependence, but also to an increased risk of suffering from mental disorders and, therefore, dual disorders.

It is therefore not an isolated or coincidental fact that both diagnosis coexist in the same individual, an affective disorder such as major depression with addiction to a substance, such as tobacco, which is called dual disorder.

In this group of patients, there is a fact worth mentioning, and that is that both diseases present an increased risk of suicidal ideation. In the case of depression, this relationship has been clearly studied, but an increased risk has also been observed in patients who are smokers or who have been smokers, which is why it is an item that has been included in different clinical scales that assess this ideation. This symptomatology requires special attention for diagnosis and treatment due to its potential lethality.

The need for new lines of treatment arises because in depression, up to 30% of patients are resistant to pharmacological therapies. Although electroconvulsive therapy is currently considered the treatment of choice for resistant depression, it has important limitations, for example due to the need to anesthetize the patient, as well as the frequent side effects that it has on cognitive functions, specifically memory loss, which make it a technique with little social acceptance. Something similar occurs with regard to nicotine use disorder. With the use of drugs such as varenicline (recently withdrawn from the market) or cytisine, the drug of choice currently for the treatment of this disorder, it is observed that only 32% of patients remain abstinent two weeks after having finished the treatment, along with the side effects that make adherence to the treatment difficult.

As a result of the therapeutic limitations described above, neuromodulation techniques, such as the one proposed in the present study: transcranial magnetic stimulation, have gained prominence in recent years.

The technique is based on Faraday's Law of electromagnetic induction. The use of a stimulation coil placed on the patient's head generates a pulse of electric current that produces a magnetic field that passes through the scalp and the cranial vault without attenuating (it only decays with the square of the distance). This magnetic pulse gives rise to a selective depolarization of neurons in the cerebral cortex, located 1.5-2 cm below the cranial vault, in such a way that it modulates their activity either by inhibiting or stimulating their effects. This entire process will depend on the shape, size, type and orientation of the coil, the strength (intensity) of the magnetic field and the frequency and duration of the transferred magnetic pulses, resulting in stimulation or inhibition of the selected areas. In addition, these changes are not restricted only to the stimulated/inhibited area, but also influence other cortical and subcortical regions through brain circuits and connections.

The FDA approved the application of the technique as a treatment for major depression in 2008. Different protocols have been approved for the treatment of this diagnosis, establishing as the main target the left dorsolateral prefrontal cortex, an area of easy accessibility for the application of the technique and which, together with others such as the cingulate region, temporal and parietal cortex regions, thalamus, hypothalamus and striatum, show hypometabolism in functional imaging tests, these alterations being, along with others, responsible for the clinical manifestations of depression.

For the treatment of tobacco addiction, the FDA approved the application of the technique in 2020, with the left dorsolateral prefrontal cortex and the insular cortex also being cortical targets. The stimulation of these two areas aims to generate changes in the mesolimbic and mesostriatal dopaminergic circuits, two regions involved in the neuropathology of addiction.

Thus, transcranial magnetic stimulation is an approved technique for the treatment of major depression and nicotine use disorder, but independently for each mental disorder. Dual disorder is also common, that is, the presence in the same patient of an addiction (nicotine) and another mental illness (major depression), and this clinical trial is proposed to evaluate the efficacy and tolerability of transcranial magnetic stimulation in patients resistant to conventional treatment, and where women are a more vulnerable group. Regarding suicidal ideation, TMS has also demonstrated its efficacy in reducing the risk in depressed patients, but not in the case of an individual with both disorders. Investigators propose this trial as an opportunity to evaluate it after applying a protocol that treats both simultaneously.

ELIGIBILITY:
Inclusion Criteria:

* Patients over 18 years of age being monitored in the mental health area of the province of Castellón, with a dual disorder: major depression and substance abuse disorder
* Patients who are refractory to two or more lines of pharmacological treatments, ensuring correct completion beforehand
* Acceptance of informed consent

Exclusion Criteria:

* Psychotic symptoms or catatonia
* Other addictions, or psychiatric or personality disorders
* Language barrier
* Mental retardation that will interfere with the ability to understand and subsequent acceptance or rejection of informed consent
* Patients diagnosed with epilepsy
* Patients diagnosed with a space-occupying lesion in the brain
* Tinnitus
* Confirmed pregnancy; if suspected, a test will be requested
* Metal piece in the body or implanted medical device, except for dental material

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-02 (Estimated); Primary Completion 2026-02 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events (Safety and Tolerability) of transcranial magnetic stimulation in the treatment of resistant major depression and smoking, in patients with dual diagnosis.. | Baseline and day 5, 10, 15 and 18. Baseline and day 108 (booster doses completed).
  The tolerability of the treatment will be measured by means of a qualitative questionnaire (YES/NO), to be filled out by the patient. The possible side effects that will be taken into account are: epileptic crisis, manic shift, syncope, transient headache, localized pain in the area of application, neck pain, paresthesia, toothache, transient changes in hearing and scalp burns.
Evaluation of the efficacy of transcranial magnetic stimulation in the treatment of resistant major depression in patients with dual disorder through the Hamilton Rating Scale. | Baseline. Baseline and day 9 and 18. Baseline and day 108 (booster doses completed).
  The effectiveness of the treatment applied will be through the evaluation of the changes produced in the affective symptoms. These changes will be evaluated with the following clinical scales:
  - Hamilton Rating Scale for Depression (HDRS). Classification of symptoms: 0 - absent; 1 - mild; 2 - moderate; 3 - severe; 4 - incapacitating. In general the higher the total score the more severe the depression. HAM-D score level of depression: 10 - 13 mild; 14-17 mild to moderate; >17 moderate to severe.
Evaluation of the efficacy of transcranial magnetic stimulation in the treatment of resistant major depression in patients with dual disorder through Clinical Global Impression Scale. | Baseline. Baseline and day 9 and 18. Baseline and day 108 (booster doses completed)
  The effectiveness of the treatment applied will be through the evaluation of the changes produced in the affective symptoms. These changes will be evaluated with the following clinical scales:
  -Clinical Global Impression (CGI) The scale consists of two sections: severity of the disease and improvement. Scores range from 1 to 7. Higher scores correspond to more severe symptoms and no improvement. A score of 0 corresponds to no evaluation.
Evaluation of the efficacy of transcranial magnetic stimulation in the treatment of resistant major depression and smoking in patients with dual disorder. | Baseline. Baseline and day 9 and 18. Baseline and 3 months (booster doses completed)
  The effectiveness of the treatment applied will be through the evaluation of the changes produced in the affective symptoms. These changes will be evaluated with the following clinical scales:
  - Montgomery-Asberg Depression Rating Scale (MADRS) It is a 10-item scale. For each item, the scale includes 7 levels of intensity/severity, scored from 0 to 6, of which 4 (0-2-4-6) are predefined and the remaining 3 (1-3-5) are reserved for intermediate situations in which it is not possible to clearly assign the degree of symptomatic intensity to any of the previous levels.
  A score below 10 points is considered to indicate the absence of depressive disorder.
Evaluation of the efficacy of transcranial magnetic stimulation in the treatment of smoking in patients with dual disorder. | Baseline. Baseline and day 9 and 18. Baseline and day 108 (booster doses completed)
  The effectiveness of the treatment applied will be through the evaluation of the changes produced in the tobacco addiction. These changes will be evaluated with the following clinical scales:
  - Fagerström test for Nicotine Dependence The scale consists of 8 items, in which scores range from 0 to 10 points. Low dependency: 0-3 Moderate dependency: 4-7 High dependency: 8-10
Evaluation of the efficacy of transcranial magnetic stimulation in the treatment of resistant major depression and smoking in patients with dual disorder. | Baseline. Baseline and day 108 (booster doses completed)
  The effectiveness of the treatment applied will be through the evaluation of the changes produced in the tobacco addiction. These changes will be evaluated with the following clinical scales:
  - Pack-year ratio calculation
Evaluation of the efficacy of transcranial magnetic stimulation in the treatment of resistant major depression and smoking in patients with dual disorder. | Baseline. Day 1,2,3,4,5,6,7,8,9,10,11,12,13,14,15,16,17 and 18. Baseline and day 108 (booster doses complete)
  The effectiveness of the treatment applied will be through the evaluation of the changes produced in the tobacco addiction. These changes will be evaluated with the following clinical scales:
  - Smoking Diary

SECONDARY OUTCOMES:
Detection by clinical scales of changes produced in different cognitive functions after treatment with transcranial magnetic stimulation in patients with dual diagnosis (resistant major depression and smoking). | Baseline. Baseline and day 9 and 18. Baseline and day 108 (booster doses completed)
  Cognitive functions will be assessed using:
  - Repeatable Battery for the Assessment of Neuropsychological Status (RBANS) The RBANS assesses immediate memory, spatial skills, language, attention, and delayed recall.
  There are no absolute values, the average is between 85 and 115. Obtaining scores below 70 will indicate significant cognitive deficits.
Detection by clinical scales of changes produced in different cognitive functions after treatment with transcranial magnetic stimulation in patients with dual diagnosis (resistant major depression and smoking). | Baseline. Baseline and day 9 and 18. Baseline and day 108 (booster doses completed)
  Cognitive functions will be assessed using:
  -Clock Drawing Test (CDT). Scores range from 10 to 0. High scores (e.g., 9-10): Generally indicate good cognitive functioning and normal task performance.
  Low scores (e.g., 3 or less): May be indicative of cognitive dysfunction
Detection by neurophysiological tests of changes produced in different cognitive functions after treatment with transcranial magnetic stimulation in patients with dual diagnosis (resistant major depression and smoking). | Baseline. Baseline and day 9 and 18. Baseline and 3 months (booster doses completed)
  Neurophysiological tests will be:
  - Cognitive potentials (P300 wave). In the P300 wave potential, the parameter evaluated is the latency at which the wave is objectified, which should be between 300-600 ms.
Detection by neurophysiological tests of changes produced in different cognitive functions after treatment with transcranial magnetic stimulation in patients with dual diagnosis (resistant major depression and smoking). | Baseline. Baseline and day 9 and 18. Baseline and day 108 (booster doses completed)
  Neurophysiological tests will be:
  - Quantified electroencephalogram (Q-EEG):
  Examination of the different frequency bands and the power of each:
  * alpha
  * beta
  * delta
  * theta

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro Fuertes, Associate Professor, Study Director — Cardenal Herrera University
Locations (1):
- Consorcio Hospitalario Provincial de Castellón, Castellon, Castellón, Spain

IPD SHARING:
Plan to Share IPD: No
The data will not publicly available due to privacy or ethical restrictions.

REFERENCES:
- [Background] Young JR, Galla JT, Appelbaum LG. Transcranial Magnetic Stimulation Treatment for Smoking Cessation: An Introduction for Primary Care Clinicians. Am J Med. 2021 Nov;134(11):1339-1343. doi: 10.1016/j.amjmed.2021.06.037. Epub 2021 Aug 15. PMID 34407423
- [Background] Prochaska JJ, Benowitz NL. Current advances in research in treatment and recovery: Nicotine addiction. Sci Adv. 2019 Oct 16;5(10):eaay9763. doi: 10.1126/sciadv.aay9763. eCollection 2019 Oct. PMID 31663029
- [Background] Posner K, Brown GK, Stanley B, Brent DA, Yershova KV, Oquendo MA, Currier GW, Melvin GA, Greenhill L, Shen S, Mann JJ. The Columbia-Suicide Severity Rating Scale: initial validity and internal consistency findings from three multisite studies with adolescents and adults. Am J Psychiatry. 2011 Dec;168(12):1266-77. doi: 10.1176/appi.ajp.2011.10111704. PMID 22193671
- [Background] Perera T, George MS, Grammer G, Janicak PG, Pascual-Leone A, Wirecki TS. The Clinical TMS Society Consensus Review and Treatment Recommendations for TMS Therapy for Major Depressive Disorder. Brain Stimul. 2016 May-Jun;9(3):336-346. doi: 10.1016/j.brs.2016.03.010. Epub 2016 Mar 16. PMID 27090022
- [Background] Mahoney JJ 3rd, Hanlon CA, Marshalek PJ, Rezai AR, Krinke L. Transcranial magnetic stimulation, deep brain stimulation, and other forms of neuromodulation for substance use disorders: Review of modalities and implications for treatment. J Neurol Sci. 2020 Nov 15;418:117149. doi: 10.1016/j.jns.2020.117149. Epub 2020 Sep 20. PMID 33002757
- [Background] Lefaucheur JP, Aleman A, Baeken C, Benninger DH, Brunelin J, Di Lazzaro V, Filipovic SR, Grefkes C, Hasan A, Hummel FC, Jaaskelainen SK, Langguth B, Leocani L, Londero A, Nardone R, Nguyen JP, Nyffeler T, Oliveira-Maia AJ, Oliviero A, Padberg F, Palm U, Paulus W, Poulet E, Quartarone A, Rachid F, Rektorova I, Rossi S, Sahlsten H, Schecklmann M, Szekely D, Ziemann U. Evidence-based guidelines on the therapeutic use of repetitive transcranial magnetic stimulation (rTMS): An update (2014-2018). Clin Neurophysiol. 2020 Feb;131(2):474-528. doi: 10.1016/j.clinph.2019.11.002. Epub 2020 Jan 1. PMID 31901449
- [Background] Kuehner C. Why is depression more common among women than among men? Lancet Psychiatry. 2017 Feb;4(2):146-158. doi: 10.1016/S2215-0366(16)30263-2. Epub 2016 Nov 15. PMID 27856392
- [Background] Koutsomitros T, Evagorou O, Schuhmann T, Zamar A, Sack AT. Advances in transcranial magnetic stimulation (TMS) and its applications in resistant depression. Psychiatriki. 2021 Dec;32(Supplement I):90-98. doi: 10.22365/jpsych.2021.054. PMID 34990384
- [Background] Ferrarelli F, Phillips ML. Examining and Modulating Neural Circuits in Psychiatric Disorders With Transcranial Magnetic Stimulation and Electroencephalography: Present Practices and Future Developments. Am J Psychiatry. 2021 May 1;178(5):400-413. doi: 10.1176/appi.ajp.2020.20071050. Epub 2021 Mar 3. PMID 33653120
- [Background] Echeverria I, Cotaina M, Jovani A, Mora R, Haro G, Benito A. Proposal for the Inclusion of Tobacco Use in Suicide Risk Scales: Results of a Meta-Analysis. Int J Environ Res Public Health. 2021 Jun 5;18(11):6103. doi: 10.3390/ijerph18116103. PMID 34198855
- [Background] Cui Y, Fang H, Bao C, Geng W, Yu F, Li X. Efficacy of Transcranial Magnetic Stimulation for Reducing Suicidal Ideation in Depression: A Meta-Analysis. Front Psychiatry. 2022 Jan 18;12:764183. doi: 10.3389/fpsyt.2021.764183. eCollection 2021. PMID 35115959
- [Background] Burke MJ, Fried PJ, Pascual-Leone A. Transcranial magnetic stimulation: Neurophysiological and clinical applications. Handb Clin Neurol. 2019;163:73-92. doi: 10.1016/B978-0-12-804281-6.00005-7. PMID 31590749
- [Background] Brini S, Brudasca NI, Hodkinson A, Kaluzinska K, Wach A, Storman D, Prokop-Dorner A, Jemiolo P, Bala MM. Efficacy and safety of transcranial magnetic stimulation for treating major depressive disorder: An umbrella review and re-analysis of published meta-analyses of randomised controlled trials. Clin Psychol Rev. 2023 Mar;100:102236. doi: 10.1016/j.cpr.2022.102236. Epub 2022 Dec 8. PMID 36587461
- See also: Related Info — https://www.who.int/es/news-room/fact-sheets/detail/depression